CLINICAL TRIAL: NCT02145832
Title: Fluconazole Versus Micafungin in Neonates With Suspected or Culture-proven Candidiasis: a Randomized Pharmacokinetic and Safety Study (TINN Project - Treat Infections iN Neonates)
Brief Title: Fluconazole Versus Micafungin in Neonates With Candidiasis
Acronym: TINN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C11-11; 2012-001916-41 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-23 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Candidiasis
Keywords: TINN; Pharmacokinetic; Neonates; Antifungal; Fluconazole; Micafungin
MeSH Terms: conditions — Candidiasis | interventions — Fluconazole; Antifungal Agents; Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluconazole (Experimental): Fluconazole Kabi, Fresenius 2mg/ml
  Fluconazole will be administered at a loading dose of 25 mg/kg on the first day and followed by a maintenance dose of 12 mg/kg or 20 mg/kg once daily, depending of corrected gestational age (GA) at the beginning of treatment:
  * 12 mg/kg/day for neonates corrected GA (GA + postnatal age) < 30 weeks
  * 20 mg/kg/day for neonates corrected GA (GA + postnatal age) ≥ 30 weeks
  The infusion will last two hours.
  Interventions: Drug: Fluconazole
- Micafungin (Experimental): Mycamine 50mg - 10 mg/mL of micafungin
  Micafungin will be administered as a loading dose of 15 mg/kg on the first day of treatment and followed by a maintenance dose of 10 mg/kg once daily.
  The infusion will last two hours.
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Fluconazole
  Other Names: Antifungal
  Arms: Fluconazole
Drug: Micafungin
  Other Names: Antifungal
  Arms: Micafungin

SUMMARY:
This study is designed to determine whether micafungin is as efficacious as the current standard of fluconazole, to compare the safety of the two drugs in the treatment of proven neonatal candidiasis.

It is also designed to further elucidate the pharmacokinetics of the two products in the growing and developing neonate and premature infant.

DETAILED DESCRIPTION:
The epidemiology of candidiasis is rapidly changing; recent estimates are that nearly 50% of Candida bloodstream isolates are non-albicans Candida species requiring the use of treatments active against them.

Because of the high risk associated with candida infection in premature babies and fluconazole prophylaxis is now recommended in Neonatal Intensive Care Units (NICUs) with a high incidence in fungal infections. As candida infection is difficult to prove and requires an urgent treatment, in particular to avoid central nervous system (CNS) infection, treatment is often started in high risk patients when the infection is only suspected, i.e. on clinical arguments without waiting for positive cultures (10% of cases).

Fluconazole has not been approved for use in the treatment of neonatal candidiasis. In contrast, the efficacy of echinocandins for the treatment of invasive candidiasis has been suggested by pre-clinical and clinical studies.

Related to Micafungin, the available data suggest that only dosages that are greater than what currently recommended in infants (2 to 4 mg/kg/day) may ensure adequate coverage of the CNS, given that ability of low dosages of micafungin to penetrate the cerebrospinal compartment and to diffuse in the cerebrospinal fluid is deemed suboptimal.

The doses that will be administered are higher that currently used in order to optimize efficacy, and the concept of a loading dose that will be used for both drugs in this project, is present in antifungal treatment strategies for adults, but it has never been applied to infants and preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates and infants between 24 up to 42 weeks gestational age AND with a post-natal age of 48 hours of life up to day of life (DOL) 120 at the time of culture acquisition.
2. Requiring antifungal therapy according to medical decision by the attending physician for microbiologically documented or clinically suspected candida infection independently from the availability of any positive culture for Candida spp
3. Written informed consent from the parents or the legally authorized representative must be obtained prior to entry.
4. Infant must have sufficient venous access to permit administration of study medication and monitoring of safety variables.
5. And specifically for the French participants: infant shall be insured (Health Insurance) - able to understand and accept the study constraints

Exclusion Criteria:

1. Infant exposed to fluconazole or micafungin prophylaxis prior to inclusion
2. Infant who has received more than 48 hours of systemic antifungal therapy (any product) prior to the first dose of study drug for treatment of the current Candida infection.
3. Infant with a concomitant medical condition, whose participation, in the opinion of the Investigator and/or medical advisor, may create an unacceptable additional risk.
4. Infant previously enrolled in this study.
5. Infant who is co-infected with a non-Candida fungal organism.
6. Neonates with isolated candiduria
7. Infant with any history of a hypersensitivity or severe vasomotor reaction to any echinocandin or fluconazole product
8. Infant with pre-existing hepatic or renal disease
9. Infants with baseline Candida spp. isolate resistant to fluconazole or micafungin according to "EUropean Committee on Antimicrobial Susceptibility Testing" and "Clinical and Laboratory Standards Institute" (EUCAST/CLSI) clinical breakpoints or with an isolate for which treatment with an alternative antifungal agent is indicated, i.e. there is insufficient evidence that the species in question is a good target for therapy with either fluconazole or micafungin.

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration / Minimal Inhibitory Concentration ratio (AUC/MIC ratio) | One year
  AUC/MIC ratio in the two treated groups (both fluconazole and micafungin) is used as primary outcome. The theoretical "Minimum Inhibitory Concentration required to inhibit the growth of 90% of organisms" (MIC90s) against the common pathogens responsible for the infection to be treated will be used by opposition with the "real MIC90" of the agent really involved that is rarely isolated.

CONTACTS AND LOCATIONS:
Locations (5):
- Antwerp, Rocourt, Liège, Louvain, Namur, Belgium
- Paris, Lyon, Saint-Pierre de La Réunion, France
- Roma, Torino, Catania, Foggia, Reggio Emilia, Italy
- Rotterdam, Amsterdam, Utrecht, Isala, Netherlands
- Malaga, Salamanca, Spain

REFERENCES:
- [Background] Leroux S, Jacqz-Aigrain E, Elie V, Legrand F, Barin-Le Guellec C, Aurich B, Biran V, Dusang B, Goudjil S, Coopman S, Garcia Sanchez R, Zhao W, Manzoni P; FP7 TINN (Treat Infections in NeoNates) consortium. Pharmacokinetics and safety of fluconazole and micafungin in neonates with systemic candidiasis: a randomized, open-label clinical trial. Br J Clin Pharmacol. 2018 Sep;84(9):1989-1999. doi: 10.1111/bcp.13628. Epub 2018 Jun 21. PMID 29744900